CLINICAL TRIAL: NCT04339972
Title: Low Intensity Focused Ultrasound Pulses (LIFUP) to Modulate Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pro00082376
Record Dates: First submitted 2020-04-01; First posted 2020-04-09 (Actual); Results first posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active LIFUP then Sham LIFUP (Experimental): Real LIFUP is delivered to the participant for visit 1, followed by sham lifup visit 2
  Interventions: Device: LIFUP
- Sham LIFUP then Active LIFUP (Sham Comparator): Sham LIFUP is delivered to the participant for visit 1, followed by real lifup visit 2
  Interventions: Device: Sham LIFUP

INTERVENTIONS:
Device: LIFUP — Low Intensity Focused Ultrasound Pulsation (LIFUP) is an interesting new form of brain stimulation that may be possible to stimulate non-invasively, safely, deep in the brain with focal precision.
  Arms: Active LIFUP then Sham LIFUP
Device: Sham LIFUP — The same as LIFUP but the device is not turned on and the subject does not receive any ultrasound.
  Arms: Sham LIFUP then Active LIFUP

SUMMARY:
The anterior nuclei of the thalamus in addition to periaqueductal gray (PAG) and rostral ventromedial medulla (RVM) are integral regions of a supraspinal opioidergic structure that regulate pain perception. With the capability to influence deep neurological tissues, low intensity frequency ultrasound pulsation (LIFUP) can likely modulate this circuit and induce analgesia. LIFUP deep brain modulation is achieved by induction of focused mechanical waveforms that traverse the cranium and underlying brain tissue. The low frequency of the ultrasonic wave consequently alters neuronal transmission and causes action potential variations through mechanical means, rather than thermal.

The purpose of this study is to examine whether stimulation of the anterior nuclei of the thalamus via LIFUP induces analgesia. We hypothesize that suppression of the anterior nuclei of the thalamus will induce a temporary increase in pain tolerance. Moreover, the behavioral changes in pain will correlate with specific regional BOLD changes during pain.

DETAILED DESCRIPTION:
LIFUP uses a single large concave, or multiple ultrasound transducers in a cap placed on the scalp to produce high frequency (100Hz) sonications for 30 seconds at a time for 10 trains of pulses. Unlike traditional diagnostic ultrasound, which constantly transmits ultrasound and 'listens' to the echo to form an image, LIFUP delivers the ultrasound in packets or pulses. For reasons that are not clear, pulsed ultrasound causes neurons to depolarize and fire. Bones typically block ultrasound waves. Cleverly, however, one can deliver the ultrasound from multiple sources and use the skull as a lens, to actually shape and focus the convergent beam deeper in the brain.

The clinical use of LIFUP thus uses MRI scans taken before stimulation to position and calculate how multiple ultrasonic pulsations will converge at a location in the brain (taking into account the bone dispersion of the beam from the skull). Since a small transducer like in diagnostic ultrasound cannot individually cause neuronal discharge, with LIFUP neuronal firing can be focused both deep (2-12cm under the cap; for comparison, traditional TMS can stimulate 1-3.4cm2 deep(9, 10)) and focally (as small as 0.5mm in diameter, and up to 1000mm; the facility of a standard, commercially-available 70mm figure-of-8 TMS coil is roughly 50mm2; (9, 10)). Interestingly, the pulse width of the carrying frequency of LIFUP (0.5ms) is strikingly similar to that used in all other pulsed neuromodulation therapies (DBS: 0.6ms, ECT: 0.5ms; TMS: 0.2ms; VNS: 0.5ms), suggesting that this timeframe is mechanistically meaningful. This is a good example of the common background science of brain stimulation that transcends the individual methods.

Researchers have examined the effects of LIFUP in preclinical and clinical settings, confirming its ability to safely stimulate neural tissue(11-14), proposing cellular mechanisms for its efficacy(13-19), and now using LIFUP in human patients(20). Monti et al. (2016) described a case study in which they used LIFUP to stimulate a comatose patient's thalamus.(20). Two pre-LIFUP assessments rated the patient as being in minimally conscious state (MCS). After sonication, the patient recovered motor and oromotor functions the next day, advancing to full language comprehension and communication by nodding and shaking his head. Five days post-LIFUP, the patient attempted to walk. While this study was neither blinded nor sham-controlled, the first application of therapeutic LIFUP in a human patient was encouraging and we expect more therapeutic applications of LIFUP and potential clinical trials in the future. If LIFUP continues to show clinical potential, it has the potential to supplant the role of DBS without the need for surgery. The key barrier to LIFUP replacing DBS for clinical applications is that by and large, DBS is used in a manner where the device is inserted and turned constantly on without attempting to fundamentally change circuit dynamics or behavior so that you could remove the device. Obviously, patients cannot permanently wear a LIFUP helmet. However, to the degree that we learn how to stimulate in ways that permanently change circuit behavior (LTD or LTP) without ablation, we may be able to substitute several sessions of LIFUP that can train and rewire the brain instead of permanently implanting hardware. LIFUP can certainly stimulate deep and focal and noninvasively and thus may be a key next step in the field of brain stimulation.

Information on the intervention to be studied. We will be using the Brainsonix Low intensity focused ultrasound pulsation device. (BX Pulsar 1001). Please see the manufacturers description (Technical Summary) along with appendixes about the actual safety of the device itself.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* Healthy volunteer

Exclusion Criteria:

* seizure history (individual or family)
* history of depression
* hospitalizations or surgeries in the previous 6 months
* currently experiencing pain
* history of chronic pain
* metal implants or objects (e.g. pacemakers, metal plates, wires)
* pregnant
* alcohol dependence
* illicit drug use in the previous 6 months
* known allergy to capsaicin
* history of brain surgery or brain lesions
* history of loss of consciousness (greater than 15 min)
* on stimulants or medications that lower seizure threshold.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
yes. After the initial data analysis is complete and the primary papers are submitted, we will release anonymized data to other credible researchers who ask.

RESULTS

PARTICIPANT FLOW:
Groups:
- Active LIFUP Followed by Sham LIFUP: Real LIFUP is delivered to the participant during this condition.
  LIFUP: Low Intensity Focused Ultrasound Pulsation (LIFUP) is an interesting new form of brain stimulation that may be possible to stimulate non-invasively, safely, deep in the brain with focal precision.
- Sham LIFUP Followed by Active LIFUP: Sham LIFUP (device turned on but no sonication delivered) during this condition
  Sham LIFUP: The same as LIFUP but the device is not turned on and the subject does not receive any ultrasound.
Period: Overall Study
Arm/Group | Active LIFUP Followed by Sham LIFUP | Sham LIFUP Followed by Active LIFUP
Started | 15 | 14
Completed | 10 | 9
Not Completed | 5 | 5
Not completed — Scheduling Issues | 3 | 3
Not completed — dropout | 1 | 1
Not completed — Technical issues | 1 | 0
Not completed — Claustraphobia | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active LIFUP Followed by Sham LIFUP | Sham LIFUP Followed by Active LIFUP | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (4.6) | 24.5 (4.6) | 24.5 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 9 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Sensory Threshold Temperature Levels (Degrees Celsius)
Description: Quantitative Sensory Testing (QST) is a valuable method for diagnosing peripheral nervous system disorders, including pain. This outcome quantifies the level of thermal stimulus temperature (degrees celsius) required for a participant to feel pain on their wrist. The temperatures will be recorded before and after LIFUP.
Time Frame: Change from Baseline 45 minutes after LIFUP in the scanner
Population: This was a crossover design so everyone in the study recieved both active and sham lifup, randomized order. Overall analysis was conducted in a repeated measure, within subject design for all 19 participants.
Measure: Mean (Standard Error); unit: Degrees Celsius
Groups:
- Active LIFUP: Real LIFUP is delivered to the participant for either visit 1 or visit 2.
- Sham LIFUP: Sham LIFUP is delivered to the participant for visit 1 or visit 2.
Arm/Group | Active LIFUP | Sham LIFUP
Number analyzed (Participants) | 19 | 19
Degrees Celsius | .51 (.3) | 1.08 (.28)

2. Primary Outcome: Number of Participants With Significant Functional MRI Blood Oxygen Level Dependent (BOLD) Signal Changes
Description: Blood oxygenation level dependent (BOLD) imaging is the standard technique used to generate images in functional MRI (fMRI) studies, and relies on regional differences in cerebral blood flow to delineate regional activity. We will measure the brain's BOLD signal as a response to thermal stimulus within the MRI scanner and determine whether a significant (p ≤ 0.005 uncorrected) increase or decrease in BOLD signal intensity is indicated as a result of either Active or Sham LIFUP.
Time Frame: Changes within 3 seconds after receiving LIFUP
Measure: Number; unit: Participants w/ significant BOLD changes
Arm/Group | Active LIFUP | Sham LIFUP
Number analyzed (Participants) | 19 | 19
Participants w/ significant BOLD changes | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: LIFUP is a safe form of brain stimulation with no risk of adverse events when administered at this intensity
Groups:
- Active LIFUP: Real LIFUP is delivered to the participant for visit 1 or visit 2.
Arm/Group | Active LIFUP | Sham LIFUP
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT04339972/Prot_SAP_000.pdf